CLINICAL TRIAL: NCT02883179
Title: Topical Lidocaine-prilocaine Cream Versus Lidocaine Infiltration for Pain Relief During Repair of Postpartum Perineal Tears: A Randomized Controlled Trial
Brief Title: Pain Relief During Repair of Postpartum Perineal Tears
Acronym: LPPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LPPT
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Improving Quality of Life
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lidocaine injection (Active Comparator): 5 mL of 2% lidocaine anhydrous solution (Depocaine) will be injected slowly along the lines of the edges of the perineal tears after delivery, with frequent aspirations to avoid intravascular injection.
  Interventions: Drug: lidocaine injection
- lidocaine-prilocaine cream (Experimental): 5-g dose of Lidocaine-prilocaine cream will be applied to the intact tissue around each tear for 5 minutes before suturing
  Interventions: Drug: lidocaine-prilocaine cream

INTERVENTIONS:
Drug: lidocaine injection — anhydrous solution
  Other Names: depocaine
  Arms: lidocaine injection
Drug: lidocaine-prilocaine cream — topical cream
  Other Names: pridocaine
  Arms: lidocaine-prilocaine cream

SUMMARY:
The aim of our study is to compare the analgesic effect of topical application of lidocaine-prilocaine cream and lidocaine infiltration during repair of postpartum perineal tears.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age > 37 weeks
2. Uncomplicated pregnancy
3. Single vertex fetus
4. Normal vaginal delivery
5. Women who will accept to participate in the study

Exclusion Criteria:

1. Women received epidural analgesia
2. Women required episiotomy
3. Women with intact perineum
4. Operative vaginal delivery
5. Allergy to the used drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Mean pain score during suture of perineal tears | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes